CLINICAL TRIAL: NCT03999619
Title: Evaluation of the Move 2 Learn (M2L) Program for Young Children: A Randomized Wait-list Controlled Trial
Brief Title: Evaluation of the Move 2 Learn (M2L) Program for Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, John Cairney, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8303
Record Dates: First submitted 2019-06-12; First posted 2019-06-26 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Motor Development; Physical Activity
Keywords: Pre-Literacy Skills
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Wait-list Controlled Design
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not be aware of the group status of children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Children will enter into the Move 2 Learn program immediately following their first assessment (between week 0 to 10)
  Interventions: Behavioral: Move 2 Learn
- Wait-list Control (Other): Children will not participate in the program until after their second assessment (between week 11 to 21). Their control period will take place between week 0 and 10.
  Interventions: Behavioral: Move 2 Learn

INTERVENTIONS:
Behavioral: Move 2 Learn — 10-week (1 hour/week) program designed to target fundamental movement and pre-literacy skills with active parent involvement.
  Other Names: M2L

SUMMARY:
Move 2 Learn (M2L) is a 10-week movement and pre-literacy program for preschool aged children and their parents designed to improve both movement and reading skills as well as support their overall cognitive, physical, and psychological development. This study will be using a randomized wait-list controlled trial design to evaluate the program on several outcomes: motor skills, pre-literacy skills, cognitive function, perceived physical competence, and physical activity. Children ages 3 to 4 years with typical development will be randomized to either start the program immediately or enter the wait-list control group to begin the program after a 10-week control period. The outcomes will be assessed for all children three times, at week 0, week 11, and week 21 to evaluate change over time in both groups.

DETAILED DESCRIPTION:
Design: The study will use a randomized wait-list controlled design. Children will be randomized to either the intervention arm or the wait-list control arm with a 1:1 ratio. Children randomized to the intervention arm will enter the Move 2 Learn (M2L) intervention during the first 10-12 weeks of the study period; children randomized to the wait-list control arm will not receive any intervention during the first 10-12 weeks of the study (the wait-list control period), then will enter into a modified M2L intervention during the second 10 to 12 weeks of the study. All children will be assessed 3 times at 10-12-week intervals. The intervention arm will be assessed before and immediately after they receive the intervention, and at a 10-12-week follow-up. The wait-list control group will be assessed at baseline, immediately before receiving the intervention (10-12 weeks following) and after they receive the intervention.

Children will be randomized 1:1 to either the intervention or wait-list control group. Simple randomization will be completed using a computer algorithm. After confirming eligibility and obtaining verbal consent, a research assistant will send the complete list of study IDs to an independent biostatistician who will use a computer algorithm to randomly assign the child to the intervention or to the wait-list control group. Sealed, opaque, and numbered envelops will be prepared with their allocation details (e.g. if randomized to the intervention arm, information regarding the location and time of the intervention will be provided).

Intervention: The Move 2 Learn (M2L) program (both the original and the modified program) will be run out of the gym space provided in-kind by the Faculty of Kinesiology and Physical Education at the University of Toronto. This behavioral program will run for 60 minutes once per week for 10 consecutive weeks and will consist of three components: direct movement skill instruction, unstructured exploratory free-play, and in interactive storybook reading activity. There is active involvement of at least one parent/caregiver in the direct instruction and reading components and parents/caregivers are provided with handouts outlining specific strategies to implement for at-home practice of the activities. Each week, parents will be verbally encouraged to practice these skills at home with their parents.

The participants randomized to the wait-list control group will not receive any intervention during the control period (between time 1 and time 2 assessments. After their time 2 assessment is complete, participants will receive a modified version of the M2L program. All in-sessions components of the M2L program will be implemented with the exception of the parent handouts and the verbal encouragement to practice at-home between sessions Assessments: At the time 1 appointment, children will be administered the gross motor subscales of the Peabody Developmental Motor Scales-2 (PDMS-2; Folio & Fewell, 2000), the perceived physical competence subscale of the Pictorial Scale (PPC) of Perceived Competence and Social Acceptance for Young Children-Preschool-Kindergarten version (PSCS-PK; Harter & Pike, 1984), the Phonological Awareness Literacy Screening: Preschool (PALS-PK; Invernizzi, Sullivan, Meier, & Swank, 2004), the Preschool Word and Print Awareness Test (PWPA; Justice & Ezell, 2002), and the Picture Deletion Task for Preschoolers (PDTP; Byrne, DeWolfe, & Bawden, 1998; Corkum, Byrne, & Ellsworth, 1995). Parents will complete a demographic questionnaire (see Demographic Survey for Parents), and a parental engagement questionnaire that asks about the use of specific activities to promote motor skill and early literacy skill development (see Parental Engagement Survey) and the Behaviour Rating Inventory of Executive Function®-Preschool Version (BRIEF-P; Gioia, Espy, & Isquith, 2001). On completion of testing, children will be fitted with an accelerometer; parents will be instructed on its proper use and provided with a diary to track wear time (e.g., time of day put on, time of day removed). After 7 days, parents will mail back the the accelerometer(s) and diary (see Accelerometer Log). At each subsequent appointment (time 2 and time 3), all outcomes described above will be measured again (see Figure 2) except for the parent demographic survey and the BRIEF-P. Each study appointment will take approximately 1.5 hours.

All outcomes will be assessed at the INfant and Child Health (INCH) Lab at the University of Toronto by trained graduate students, blind to the intervention status of the participants.

Measures: The primary outcomes include fundamental movement skills and pre-literacy skills. Movement skills will be assessed using the gross motor sub-scales of the Peabody Developmental Motor Scales - 2 (PDMS-2). The Preschool Word and Print Awareness Test (PWPA) and the Phonological Awareness Literacy Screening: Preschool (PALS-PK) to measure print-concept knowledge and alphabet knowledge, respectively. Secondary outcomes include physical activity, cognitive function, and self-perceived physical competence. All outcomes will be assessed at the INfant and Child Health (INCH) Lab at the University of Toronto by trained graduate students, blind to the intervention status of the participants.

Motor Skill Proficiency: The gross motor subscales of the PDMS-2 (stationary performances, locomotion, and object manipulation) will be used to assess change in motor skill over the course of the study and will be administered by a trained graduate student blind to the intervention status of the participant. This tool is commercially available.

Pre-literacy Skills: Emergent literacy skills that will be measured include print concepts and alphabet knowledge. The PALS-PK Upper-case Alphabet Recognition task will be used to measure children's alphabet knowledge. This tool is commercially available. Print awareness will be assessed using the PWPA. The assessment uses an interactive story book reading activity to test children on their knowledge of 14 print concepts, such as print directionality and print function (Justice & Ezell, 2002). This tool is freely available as it was published as an appendix in the Justice, Bowles, & Skibbe, 2006 article.

Physical Activity: Accelerometry is an objective method of assessing free-moving physical activity, and is the method best-suited to measuring activity in young children. This study will use the Actigraph GT3X activity monitor, a light (27g) and small (3.8cm × 3.7cm × 1.8cm) device, secured to the child by a belt worn around the waist. A 3 s epoch will be used (Obeid, Nguyen, Gabel, & Timmons, 2011) and will record physical activity for 7 consecutive days (Trost, Pate, Freedson, Sallis, & Taylor, 2000).

Executive Function: The BRIEF-P, a parent-report tool, will be used to assess children's trait executive function at week 0 (Sherman & Brooks, 2010). State executive function will be assessed using the Attention Sustained subtest 6 of the Leiter-3 test battery. The task requires children to view a target image (an animal) and identify the images that match among a set of distractor images as quickly as possible; there are 4 trials, each of which have a practice set. This tool is commercially available. To assess inhibition, the Head Toes Knees and Shoulders instrument will also be administered. This task requires Children are to play a game in which they must do the opposite of what the experimenter says. The experimenter instructs children to touch their head (or their toes), but instead of following the command, the children are supposed to do the opposite and touch their toes.

Perceived Physical Competence: The PSCS-PK will be used to assess each child's level of perceived competence. There are physical competence subscale (6-items) will be administered. The scale is an extension of Harter's Perceived Competence Scale for Children (1982). This tool is freely available online.

Demographic Factors: The baseline questionnaire will include questions about the parent and the child on age, gender, race/ethnicity, parental education and occupation, and household income. The questionnaire will be parent-completed.

Parental Engagement: Parents will be asked about the use and the frequency of use, of specific activities that will be employed in our program. A parent-reported questionnaire specific to these activities has been created to determine if parents have been using these strategies before our program, and if they have incorporated them into their activities with their child after having completed the program.

Parental Acceptability: Consenting parents will engage in a focus group, led by a facilitator. Staying consistent with the unstructured nature of a focus group, open-ended questions designed to initiate discussions surrounding their attitudes and opinions, likes and dislikes of the program will be asked. The discussion will be audio recorded and transcribed verbatim. Focus group transcriptions will be used to revise the program and its components to better serve the community.

Analysis: Basic descriptive statistics of participating children and parents will be completed. Mixed effects models will be used to assess a group-by-time effect on all outcomes. All analyses will be conducted on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 3 and 4 years with typical development

Exclusion Criteria:

* Developmental delay
* Physical conditions that prohibit safe participation in physical activity

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Motor skills | Change from week 0 to 11
  Movement skill competency (Peabody Developmental Motor Scales- 2nd ed; total gross motor scores range from 0 to 286 with higher scores representing higher motor skill)
Change in Pre-literacy skills | Change from week 0 to 11
  Print Concept Knowledge (Preschool Word and Print Awareness Tool; standardized scores range from 0 to 181 with higher scores representing higher pre-literacy skill)

SECONDARY OUTCOMES:
Change in Perceived Physical Competence | Change from week 0 to 11
  Perceptions of one's own physical abilities (Physical Competence subscale of Harter's Pictorial Scale of Perceived Competence and Social Acceptance for Young Children; subscale scores range from 4 to 24 and will be averaged to produce a score ranging from 1 to 4 with higher scores representing more positive self perceptions)
Change in Perceived Physical Competence | Change from week 11 to 21
  Perceptions of one's own physical abilities (Physical Competence subscale of Harter's Pictorial Scale of Perceived Competence and Social Acceptance for Young Children; subscale scores range from 4 to 24 and will be averaged to produce a score ranging from 1 to 4 with higher scores representing more positive self perceptions)
Change in Executive function - Attention | Change from week 0 to 11
  Sustained Attention (Subtest 6 of the Leiter-3; scores of correct responses range from 0 to 70 with high scores representing higher levels of attention; scores of errors of commission range from 0 to 205 with higher scores representing lower levels attention)
Change in Executive function - Attention | Change from week 11 to 21
  Sustained Attention (Subtest 6 of the Leiter-3; scores of correct response range from 0 to 70 with high scores representing higher levels of attention; scores of errors of commission range from 0 to 205 with higher scores representing lower levels of attention)
Executive function - Inhibition | Change from week 0 to 11
  Inhibition (Head Toes Knees Shoulders Instrument; scores range from 0 to 52 with higher score representing higher inhibition)
Executive function - Inhibition | Change from week 11 to 21
  Inhibition (Head Toes Knees Shoulders Instrument; scores range from 0 to 52 with higher score representing higher inhibition)
Physical activity | Change from week 0 to 11
  Levels of physical activity over 7 days as measured using accelerometers
Physical activity | Change from week 11 to 21
  Levels of physical activity over 7 days as measured using accelerometers
Parental engagement - movement activity | Change from week 0 to 11
  Parent-reported levels of engagement in completing movement activities at home
Parental engagement - movement activity | Change from week 11 to 21
  Parent-reported levels of engagement in completing movement activities at home
Parental engagement - reading activity | Change from week 0 to 11
  Parent-reported levels of engagement in completing pre-literacy activities at home
Parental engagement - reading activity | Change from week 11 to 21
  Parent-reported levels of engagement in completing pre-literacy activities at home
Change in Motor skills | Change from week 11 to 21
  Movement skill competency (Peabody Developmental Motor Scales- 2nd ed; total gross motor scores range from 0 to 286 with higher scores representing higher motor skill)
Change in Pre-literacy skills | Change from week 11 to 21
  Print Concept Knowledge (Preschool Word and Print Awareness Tool; standardized scores range from 0 to 181 with higher scores representing higher pre-literacy skill)

CONTACTS AND LOCATIONS:
Overall Officials: John Cairney, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No